CLINICAL TRIAL: NCT03187769
Title: A Study to Evaluate the Effect of ALKS 3831 Compared to Olanzapine on Body Weight in Young Adults With Schizophrenia, Schizophreniform, or Bipolar I Disorder Who Are Early in Their Illness
Brief Title: Study to Evaluate the Efficacy of ALKS 3831 on Body Weight in Young Adults Who Have Been Recently Diagnosed With Schizophrenia, Schizophreniform, or Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALKS 3831-A307
Record Dates: First submitted 2017-06-08; First posted 2017-06-15 (Actual); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Schizophrenia; Schizophreniform Disorders; Bipolar I Disorder
Keywords: Alkermes; ALKS 3831; Olanzapine; Samidorphan; Schizophrenia; Schizophreniform; Bipolar I
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALKS 3831 (Experimental): Coated bilayer tablet
  Interventions: Drug: ALKS 3831
- Olanzapine (Active Comparator): Coated bilayer tablet
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: ALKS 3831 — Olanzapine + samidorphan, daily oral dosing
  Arms: ALKS 3831
Drug: Olanzapine — Daily oral dosing
  Arms: Olanzapine

SUMMARY:
This study will evaluate the effect of ALKS 3831 compared to olanzapine on body weight in young adults with schizophrenia, schizophreniform, or bipolar I disorder who are early in their illness

DETAILED DESCRIPTION:
In the US adolescent subjects starting at age 16 will be enrolled. In the EU, subjects age 18 and older will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Has less than 24 weeks previous treatment with antipsychotics (cumulative; lifetime)

  * Subject treated with aripiprazole can receive an additional 1 year of treatment at ≤5 mg/day, and this treatment will not be considered as part of the 24 weeks of previous treatment with antipsychotics
* Has less than 4 years elapse since the initial onset of active-phase of symptoms
* Has a body mass index (BMI) of <30 kg/m^2
* Agrees to use an acceptable method of contraception for the duration of the study and for 30 days after the last dose of study drug
* Subject meets the criteria for a primary diagnosis of schizophrenia, schizophreniform disorder, or bipolar I disorder
* For bipolar I disorder, must have been experiencing an episode of acute mania within ≤14 days prior to Visit 1
* Suitable for outpatient treatment
* Additional criteria may apply

Exclusion Criteria:

* Poses a current suicide risk
* Has a history of poor or inadequate response to treatment with olanzapine
* Has previously been treated with long-acting injectable antipsychotic medication within the 2 months prior to screening, or has > 6 months cumulative life use, or has received treatment with electroconvulsive therapy in their lifetime
* Has initiated treatment with mood stabilizers (eg lithium, valproate, etc) >2 months prior to Visit 1
* Has a positive drug screen for opioids, phencyclidine (PCP), amphetamine/methamphetamine, or cocaine
* Has taken opioid agonists (eg, codeine, oxycodone, tramadol, morphine) within the 14 days prior to Visit 1, or has taken opioid antagonists, including naltrexone and naloxone, within 60 days prior to Visit 1
* Taking any weight loss agents or hypoglycemic agents
* Has a clinically significant or unstable medical illness, condition, or disorder that would be anticipated to potentially compromise subject safety or adversely affect the evaluation of efficacy
* Has joined a weight management program or had significant changes in diet or exercise regimen within the past 6 weeks
* Has started a smoking cessation program within the past 6 months
* Has a history of diabetes
* Currently pregnant or breastfeeding or is planning to become pregnant during the study or within 30 days of the last study drug administration
* Additional criteria may apply

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 426 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkermes Medical Director, Study Director — Alkermes, Inc.
Locations (54):
- United States (22):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Rogers, Arkansas
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, San Diego, California
  - Alkermes Investigational Site, Stanford, California
  - Alkermes Investigational Site, Jacksonville, Florida
  - Alkermes Investigational Site, North Miami, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Augusta, Georgia
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Winfield, Illinois
  - Alkermes Investigational Site, Kalamazoo, Michigan
  - Alkermes Investigational Site, Kansas City, Missouri
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Las Vegas, Nevada
  - Alkermes Investigational Site, Cincinnati, Ohio
  - Alkermes Investigational Site, Eugene, Oregon
  - Alkermes Investigational Site, DeSoto, Texas
  - Alkermes Investigational Site, Fort Worth, Texas
  - Alkermes Investigational Site, Houston, Texas
  - Alkermes Investigational Site, Richardson, Texas
  - Alkermes Investigational Site, San Antonio, Texas
- Alkermes Investigational Site, Vienna, Austria
- Alkermes Investigational Site, München, Germany
- Alkermes Investigational Site, Galway, Ireland
- Israel (2):
  - Alkermes Investigational Site, Jerusalem
  - Alkermes Investigational Site, Tel Litwinsky
- Italy (3):
  - Alkermes Investigational Site, Brescia
  - Alkermes Investigational Site, Naples
  - Alkermes Investigational Site, Torino
- Alkermes Investigational Site, Poznan, Poland
- Russia (8):
  - Alkermes Investigational Site, Arkhangelsk
  - Alkermes Investigational Site, Moscow
  - Alkermes Investigational Site, Roshchino
  - Alkermes Investigational Site, Rostov-on-Don
  - Alkermes Investigational Site, Saint Petersburg
  - Alkermes Investigational Site, Samara
  - Alkermes Investigational Site, Saratov
  - Alkermes Investigational Site, Tonnel’nyy
- South Korea (4):
  - Alkermes Investigational Site, Busan
  - Alkermes Investigational Site, Daegu
  - Alkermes Investigational Site, Naju
  - Alkermes Investigational Site, Seoul
- Alkermes Investigational Site, Oviedo, Spain
- Ukraine (6):
  - Alkermes Investigational Site, Kharkiv
  - Alkermes Investigational Site, Kyiv
  - Alkermes Investigational Site, Lviv
  - Alkermes Investigational Site, Poltava
  - Alkermes Investigational Site, Smila
  - Alkermes Investigational Site, Stepanovka
- United Kingdom (4):
  - Alkermes Investigational Site, Guildford
  - Alkermes Investigational Site, Headington
  - Alkermes Investigational Site, London
  - Alkermes Investigational Site, Maidstone

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kahn RS, Kane JM, Correll CU, Arevalo C, Simmons A, Graham C, Yagoda S, Hu B, McDonnell D. Olanzapine/Samidorphan in Young Adults With Schizophrenia, Schizophreniform Disorder, or Bipolar I Disorder Who Are Early in Their Illness: Results of the Randomized, Controlled ENLIGHTEN-Early Study. J Clin Psychiatry. 2023 Mar 22;84(3):22m14674. doi: 10.4088/JCP.22m14674. PMID 36946605

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ALKS 3831 | Olanzapine
Started | 211 | 215
Completed | 165 | 161
Not Completed | 46 | 54

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all randomized subjects who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | ALKS 3831 | Olanzapine | Total
Number analyzed (Participants) | 211 | 215 | 426
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (6.12) | 25.7 (5.92) | 25.8 (24.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 75 | 144
  Male | 142 | 140 | 282
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 14 | 26
  Not Hispanic or Latino | 199 | 201 | 400
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 3 | 10 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 62 | 58 | 120
  White | 139 | 144 | 283
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Austria | 0 | 2 | 2
  South Korea | 0 | 2 | 2
  United States | 102 | 104 | 206
  Ireland | 1 | 3 | 4
  Ukraine | 35 | 42 | 77
  Poland | 1 | 1 | 2
  Italy | 9 | 4 | 13
  United Kingdom | 2 | 1 | 3
  Israel | 20 | 12 | 32
  Germany | 1 | 2 | 3
  Russia | 40 | 42 | 82
Weight [Mean (Standard Deviation); unit: Kilogram (kg)] — Kilogram (kg)
  Kilogram (kg) | 71.57 (13.278) | 70.09 (12.366) | 70.83 (12.832)
Clinical Global Impression-Severity (CGI-S) Score [Mean (Standard Deviation); unit: units on a scale] — The CGI-S is a 7-point scale that requires the clinician to assess how mentally ill the patient is at a specific point in time. Based on the scale, patients are categorized as follows: "1: normal, not at all ill"; "2: borderline mentally ill"; "3: mildly ill"; "4: moderately ill"; "5: markedly ill"; "6: severely ill"; and "7: among the most extremely ill patients." Population: The Full Analysis Set (FAS) includes all subjects in the Safety Population who have at least 1 post-baseline weight assessment.
  For the secondary efficacy endpoint, the LS mean (±SE [95% CI]) change from baseline in CGI S score was measured within the ALKS 3831 Group at Week 12.
  units on a scale
    number analyzed (Participants) | 202 | 0 | 202
    (all) | 3.87 (.809) |  | 3.87 (.809)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Weight at Week 12
Description: The efficacy analyses were performed using the Final Analysis Set which is defined as all randomized subjects who received one dose of study drug and had at least 1 primary efficacy assessment after administration of study drug
Time Frame: Baseline and 12 weeks
Population: The efficacy analyses were performed using the Final Analysis Set (FAS) which is defined as all randomized subjects who received one dose of study drug and had at least 1 primary efficacy assessment after administration of study drug
Measure: Least Squares Mean (Standard Error); unit: Percentage of change in body weight
Arm/Group | ALKS 3831 | Olanzapine
Number analyzed (Participants) | 202 | 206
Percentage of change in body weight | 4.91 (.597) | 6.77 (.596)
Statistical Analysis 1: Comparison: ALKS 3831; Test type: Superiority; p = .012, ANCOVA; Least Squares Mean Difference = -1.87, 95% CI 2-sided [-3.33 to -.41]

2. Secondary Outcome: Percentage of Subjects With ≥10% Weight Gain at Week 12
Description: Percentage of weight gain is analyzed based on the subject's assessment status (≥10% vs <10%) at Week 12 using a logistic regression model including treatment group, diagnosis (schizophrenia/schizophreniform disorder vs bipolar I disorder), region (US vs non-US), and baseline BMI (<25 vs ≥25) as factors and baseline weight as covariate.
Time Frame: Baseline and 12 weeks
Population: The efficacy analyses were performed using the Final Analysis Set which is defined as all randomized subjects who received one dose of study drug and had at least 1 primary efficacy assessment after administration of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | ALKS 3831 | Olanzapine
Number analyzed (Participants) | 202 | 206
Percentage of participants | 21.9 | 30.4

3. Secondary Outcome: Percentage of Subjects With ≥7% Weight Gain at Week 12
Time Frame: Baseline and 12 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ALKS 3831 | Olanzapine
Number analyzed (Participants) | 202 | 206
Percentage of participants | 33.1 | 44.8

4. Secondary Outcome: Number of Participants Experiencing of Adverse Events (AEs)
Time Frame: Up to 16 weeks
Population: The safety population included all subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ALKS 3831 | Olanzapine
Number analyzed (Participants) | 211 | 215
Participants | 134 | 136

5. Secondary Outcome: Change From Baseline in Waist Circumference at Week 12
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Centimeters
Arm/Group | ALKS 3831 | Olanzapine
Number analyzed (Participants) | 202 | 206
Centimeters | 2.99 (.464) | 3.90 (.477)

6. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score Within the ALKS 3831 Group at Week 12
Description: Clinical Global Impression-Severity (CGI-S) Score is a 3-item, clinician-rated scale used to assess global illness severity, overall improvement from the start of treatment, and therapeutic response. It is a 7-point scale that requires the clinician to assess how mentally ill the patient is at a specific point in time. Based on the scale, patients are categorized as follows: "1: normal, not at all ill"; "2: borderline mentally ill"; "3: mildly ill"; "4: moderately ill"; "5: markedly ill"; "6: severely ill"; and "7: among the most extremely ill patients."
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ALKS 3831
Number analyzed (Participants) | 202
units on a scale | -.82 (.060)

ADVERSE EVENTS:
Time Frame: 16 Weeks
Arm/Group | ALKS 3831 | Olanzapine
All-Cause Mortality (participants affected / at risk) | 1/211 | 0/215
Serious Adverse Events (participants affected / at risk) | 8/211 | 8/215
Other Adverse Events (participants affected / at risk) | 134/211 | 136/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALKS 3831 (N=211) | Olanzapine (N=215)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 2
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 2
Seizure (Nervous system disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Varicella (Infections and infestations) | 1 | 0
Limb deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 3 | 2
Bipolar I Disorder (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALKS 3831 (N=211) | Olanzapine (N=215)
Weight Increased (Investigations) | 46 | 55
Somnolence (Nervous system disorders) | 23 | 20
Alanine aminotransferase increased (Investigations) | 16 | 14
Headache (Nervous system disorders) | 13 | 10
Sedation (Nervous system disorders) | 11 | 13
Waist Circumference Increased (Investigations) | 10 | 15
Nausea (Gastrointestinal disorders) | 9 | 5
Anxiety (Psychiatric disorders) | 8 | 12
Blood creatine phosphokinase increased (Investigations) | 8 | 5
Fatigue (General disorders) | 8 | 4
Aspartate aminotransferase increased (Investigations) | 7 | 8
Dizziness (Nervous system disorders) | 6 | 3
Dry mouth (Gastrointestinal disorders) | 6 | 1
Increased appetite (Metabolism and nutrition disorders) | 6 | 9
Vomiting (Gastrointestinal disorders) | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.

DOCUMENTS (2):
  • Study Protocol (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT03187769/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/69/NCT03187769/SAP_001.pdf